CLINICAL TRIAL: NCT01471210
Title: A Phase 1 Study of the Safety, Tolerability, Pharmacokinetics and Immunoregulatory Activity of Urelumab (BMS-663513) in Subjects With Advanced and/or Metastatic Solid Tumors and Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma (B-NHL)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Immunoregulatory Study of Urelumab (BMS-663513) in Subjects With Advanced and/or Metastatic Solid Tumors and Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA186-011; 2012-000170-28 (EudraCT Number)
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2016-08

CONDITIONS: Cancer - Solid Tumors and B-Cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 : Urelumab (BMS-663513) Dose escalation (Experimental): Urelumab (BMS-663513) solution administered intravenously on specified days
  Interventions: Drug: Urelumab (BMS-663513)
- Part 2 : Urelumab (BMS-663513) Cohort Expansion (Experimental): Urelumab (BMS-663513) solution administered intravenously on specified days
  Interventions: Drug: Urelumab (BMS-663513)
- Part 3:Urelumab (BMS-663513) Tumor-specific Cohort Expansions (Experimental): Enrollment of subjects of three specific tumor types [(colorectal cancer (CRC), head and neck squamous cell carcinoma (SCCHN), and B-Cell non-Hodgkin's lymphoma (B-NHL)] who will be treated at the Maximum Tolerated Dose (MTD) (or highest dose tested)
  Interventions: Drug: Urelumab (BMS-663513)
- Part 4:Urelumab (BMS-663513) Cohort Expansion in B-NHL (Experimental): Arm A and Arm B: Urelumab (BMS-663513) liquid administered intravenously on specified days exploring q3w and q6w dosing regimen
  Interventions: Drug: Urelumab (BMS-663513)

INTERVENTIONS:
Drug: Urelumab (BMS-663513)

SUMMARY:
The purpose of the study is to assess the safety, tolerability, pharmacokinetics and immunoregulatory activity of urelumab (BMS-663513) in cancer subjects with advanced and/or metastatic tumors and relapsed/refractory B-Cell Non-Hodgkin's Lymphoma

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

1. Signed Written Informed Consent

   * The signed informed consent form
2. Target Population

   * Subjects with advanced and/or metastatic solid tumors or B-NHL who are either refractory to or have relapsed from standard therapies, or for whom a standard therapy does not exist with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
   * Life expectancy of 12 weeks or greater
   * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
   * Adequate organ and marrow function
   * For certain subjects, willing and able to provide pre- and post-treatment fresh tumor biopsies
3. Age and Reproductive Status

   * Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy throughout the study and for at least 4 weeks prior to initiation of dosing, and for at least 60 days after the last dose of investigational product in such a manner that the risk of pregnancy is minimized
   * WOCBP must have a negative serum or urine pregnancy test [minimum sensitivity 25 UI/L or equivalent units of human chorionic gonadotrophin (HCG)] within 24 hours prior to the start of investigational product
   * Women must not be breastfeeding

Exclusion Criteria:

1. Target Disease Exceptions

   * Subjects with known or suspected brain metastasis unless previously treated and without evidence of progression
   * Subjects with a history of prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured
   * Subjects with hepatocellular carcinoma
2. Medical History and Concurrent Diseases

   * Any active autoimmune disease or documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo, psoriasis inactive within past 2 years, resolved childhood asthma/atopy, or thyroid disease controlled by replacement therapy without the need for immunosuppression
   * Known or suspected human immunodeficiency virus (HIV) or hepatitis A(acute), B or C infection
   * History of any hepatitis (e.g., alcohol or non-alcohol steatohepatitis (NASH), drug-related, auto-immune)
   * Evidence of active infection, requiring parenteral anti-bacterial, anti-viral or anti-fungal therapy < 7 days prior to administration of study medication
   * History of clinically significant cardiac disease, including but not limited to a history (personal or family) of congenital long QT syndrome
   * Grade > 1 QTc prolongation at baseline (> 450 msec by Bazett formula) confirmed by a repeat electrocardiogram (ECG)
   * History of myocardial infarction or uncontrolled angina within 12 months prior to administration of study drug
3. Physical and Laboratory Test Findings

   * WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 12 weeks after the last dose of investigational product
   * Women who are pregnant or breastfeeding
   * Women with a positive pregnancy test on enrollment or prior to investigational product administration
   * Sexually active fertile men not using effective birth control if their partners are WOCBP
   * Positive blood screen for hepatitis A IgM, hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody
4. Allergies and Adverse Drug Reaction

   * History of allergy to Urelumab (BMS-663513) or related compounds
   * History of significant drug allergy (such as anaphylaxis or hepatotoxicity) to a prior biologic therapy
5. Prohibited Treatments and/or Therapies

   * The systemic use of the following therapies are prohibited within 28 days of first dose of study medication, or longer where indicated:

     1. Use of anti-cancer treatment (including investigational drugs) within 28 days
     2. Immunosuppressive medications or immunosuppressive doses of systemic corticosteroids
     3. Surgery (except minor surgeries,e.g., biopsies) or radiotherapy
     4. Any non-oncology live viral vaccine therapies used for the prevention of infectious diseases.
   * Prior treatment with anti-programmed death 1 (anti-PD-1)/Programmed cell death 1 ligand 1 (PD-L1) or anti-CD137
   * Any subject with the following reported drug-related adverse events on anti- Cytotoxic T-Lymphocyte Antigen 4 (anti-CTLA4) will not be permitted on study: hepatic, diarrhea/colitis or endocrine adverse events (AE)s Grade ≥ 2, any other non-laboratory immune-related AE ≥ Grade 3. Subjects must have minimum 9 week washout period between the last dose of anti-CTLA4 and the first dose Urelumab (BMS-663513)
   * Prior organ allograft or allogeneic bone marrow transplantation
6. Other Exclusion Criteria

   * Prisoners or subjects who are involuntarily incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, physical examinations, and clinical laboratory tests | Every 3 weeks from Baseline (Day 1) for up to 2 years
  The incidence of adverse events will be tabulated and reviewed for potential significance and clinical Importance.
Dose-limiting toxicity and maximum tolerated dose of Urelumab (BMS-663513) as determined by the incidence of dose-limiting toxicities | Every 3 weeks from Baseline (Day 1) for up to 9 weeks of therapy

SECONDARY OUTCOMES:
Maximum observed serum concentrations (Cmax) of Urelumab (BMS-663513) | Cycle 1 Day 1
Minimum observed serum concentrations (Cmin) of Urelumab (BMS-663513) | Cycle 2 Day 1, Cycle 3 Day 1, every 12 weeks thereafter up to 2 years
Time of maximum observed serum concentration (Tmax) of Urelumab (BMS-663513) | Cycle 1 Day 1
Area under the concentration-time curve in 1 dosing interval [AUC(TAU)] of Urelumab (BMS-663513) | Cycle 1 Day 1 - Day 4, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 3 Day 1 and every 12 weeks thereafter up to 2 years
Plasma half-life (T-HALF) of Urelumab (BMS-663513) | Cycle 1 Day 1 - Day 4, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 3 Day 1 and every 12 weeks thereafter up to 2 years
Total body clearance (CLT) of Urelumab (BMS-663513) | Cycle 1 Day 1 - Day 4, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 3 Day 1 and every 12 weeks thereafter up to 2 years
Volume of distribution at steady-state (Vss) of Urelumab (BMS-663513) | Cycle 1 Day 1 - Day 4, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 3 Day 1 and every 12 weeks thereafter up to 2 years
Human Anti-human Antibodies | Cycle 1 Day 1 - Day 4, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 3 Day 1 and every 12 weeks thereafter up to 2 years
  Immunogenicity of Urelumab (BMS-663513), as determined by blood sample measurements of human antihuman antibodies (HAHA)
Tumor response and progression as determined by proportion of patients with best overall response (BOR), progression-free survival (PFS), objective response rate (ORR), time to response, and duration of response | 9 weeks from Baseline (Day 1) and every 9 weeks until disease progression, death or last tumor assessment (Approximately up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (12):
  - Division Of Hematology & Oncology Ctr. For Health Sciences, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University Of Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Portland Med Ctr, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - University Of Virginia Health System, Charlottesville, Virginia
- France (8):
  - Local Institution, Créteil
  - Local Institution, Lille
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Pierre-Bénite
  - Local Institution, Rennes
  - Local Institution, Rouen
  - Local Institution, Villejuif
- Local Institution, Essen, Germany
- Spain (3):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Local Institution, Pamplona

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx